CLINICAL TRIAL: NCT04401566
Title: Investigation of Acute Effects of Myofascial Trigger Point Release Techniques Using Transperineal Ultrasound in Women With Chronic Pelvic Pain
Brief Title: Investigation of Acute Effects of Myofascial Trigger Point Release in Women With Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Alime Buyuk, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: :60116787-020/47015
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Pelvic Pain; Pelvic Floor; Relaxation; Myofascial Trigger Point Pain
Keywords: pelvic pain; myofascial trigger point release; transperineal ultrasound
MeSH Terms: conditions — Pelvic Pain; Myofascial Pain Syndromes | interventions — Control Groups

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The gynecologist was blind about treatment and the investigator was blind about assesment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internal Myofascial Release Group (Experimental): Internal myofascial trigger point release therapy consists of 30 minutes massage directly to the pelvic floor musculature by vaginally. Patients were instructed in internal myofascial release techniques. Experienced pelvic health physiotherapist (A.B.) to use her fingers with a lubricated glove when the finger could easily reach internal trigger points and follows these steps: (a) finding internal and external trigger points associated with pelvic muscles, especially around sensitive areas of the vagina, anus, and/or pelvic floor; (b) releasing with the fingers the trigger point associated pelvic muscle tension by carefully pressing on the trigger point. Releasing pelvic muscle tension includes applying varying amounts of pressure, sometimes gradually stroking and strumming the muscle region while systematically contracting and relaxing the affected muscles to aid in a trigger point release.
  Interventions: Other: Internal myofascial release
- External Myofascial Release Group (Experimental): Eksternal myofascial trigger point release therapy consists of 30 minutes massage to the abdominal wall, gluteal area and abductors, and hamstring muscles. Pain in trigger points may exist at both locations of muscle insertion as well as in the belly and the lower extremity of the muscle.
  Interventions: Other: External myofascial release
- Control Group (Other): The Control group will have a video about exercises recommended in pelvic pain for 30 minutes. A physiotherapist will teach and show the exercises for pelvic pain. The home exercise for pelvic pain contains diaphragm breathing, pelvic floor muscle stretching, and releasing.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Internal myofascial release — Internal myofascial trigger point release therapy consist of 30 minutes massage directly to the pelvic floor musculature by vaginally. Patients were instructed in internal myofascial relase techniques. Experienced pelvic health physiotherapist (A.B.) to use her fingers with a lubricated glove when the finger could easily reach internal trigger points and follows these steps: (a) finding internal and external trigger points associated with pelvic muscles, especially around sensitive areas of the vagina, anus, and/or pelvic floor; (b) releasing with the fingers the trigger point associated pelvic muscle tension by carefully pressing on the trigger point
  Arms: Internal Myofascial Release Group
Other: External myofascial release — Eksternal myofascial trigger point release therapy consist 30 minutes massage to the abdominal wall, gluteal area and adductors and hamstring muscles. Pain in trigger points may exist at both locations of muscle insertion as well as in the belly and lower extremity of the muscle.
  Arms: External Myofascial Release Group
Other: Control Group — The Control group will have a paper about exercises recommended in pelvic pain for 30 minutes. A physiotherapist will teach and show the exercises for pelvic pain. The home exercise for pelvic pain contains diaphragm breating, pelvic floor muscle stretching and releasing.
  Arms: Control Group

SUMMARY:
The patients diagnosed with pelvic pain will be included in the study. Orthopedic tests for pelvic pain were performed after routine gynecological examinations. After perineometer measurement, pelvic floor muscle sensitivity grading, ultrasound, and pain score evaluation, participants will be randomized and divided into 3 groups. According to a randomization plan the first group will be instructed by a physiotherapist to receive an internal myofascial trigger point release technique, the second group receive an external myofascial trigger point release technique, and the third group receive a video of relaxation exercises related to pelvic pain. After the application, measurement of perineometer and pelvic floor muscle sensitivity grading, ultrasound, and pain evaluations will be repeated.

DETAILED DESCRIPTION:
Turkey has been affected country from a busy and stressful lifestyle in our changing world and that leads to pelvic floor dysfunction has increased rapidly in Turkey. Pelvic pain that has in 1 out of every 7 women causes overactivity of pelvic floor muscles with increasing stress factors. In addition, it becomes chronic due to both the diagnosis process and the time-out of the right treatment and deteriorates the quality of life of women. There is no special pelvic floor physiotherapy for the management of pelvic pain in our country, which also causes psychosocial problems. On the other hand, myofascial trigger point release technique, which is proposed in addition to medical treatment alone or in pelvic floor physiotherapy, has been one of the current research areas in the world. However, there is no study in the national and international literature comparing internal and external myofascial trigger point relaxation techniques and also evaluating transperineal ultrasound. This study is unique in terms of comparing two different applications (internal and external trigger point relaxation technique) with ultrasound measurements in the literature.

33 women diagnosed with pelvic pain between the ages of 18-55 will be included in this study. Orthopedic tests for pelvic pain will be performed after routine gynecological examinations. After perineometer measurement, pelvic floor muscle sensitivity grading, ultrasound and pain score evaluation, participants will be randomized and divided into 3 groups. The first group will receive internal myofascial trigger point release technique, the second group will receive external myofascial trigger point release technique, and the third group will be shown a video of relaxation exercises related to pelvic pain. After the application, measurement of perineometer and pelvic floor muscle sensitivity grading, ultrasound and pain evaluations will be repeated.

ELIGIBILITY:
The inclusion criteria:

* to have chronic pelvic pain for more than six months,
* to have 5 pelvic pain orthopedic tests (active straight leg raise (ASLR), flexion abduction external rotation (FABER), pelvic pain provocation (P4), long dorsal ligament palpation (LDL), The Gaenslen Test) and at least three of the tests are positive,
* to have good communication skills and accept to attend the study.

The exclusion criteria:

* pregnant women who have had a pregnancy in the last year or who are breastfeeding;
* other causes of pain (eg pain unrelated to pelvic region relations, dermatological conditions, herpes, vulvovaginal atrophy);
* menopause;
* urogynecological conditions (i.e. pelvic prolapse grade >3 according to the Pelvic Organ Prolapse - Quantification method (POP-Q) or a urinary or vaginal infection active or present in the last 3 months);
* history of pelvic floor surgery (e.g. corrective surgery for organ descent, urinary incontinence, hysterectomy, mesh surgery,TVT,TOT);
* previous pelvic floor rehabilitation treatments; 7) expected changes in medication that may affect the perception of pain (eg pain relievers, antidepressants);
* any other medical conditions that may interfere with the study procedures (eg hormonal, psychological, cardiovascular, hematological, neurological, pulmonary or renal);
* refusal to abstain from other treatments until the end of their participation in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2021-05-02 (Actual)

PRIMARY OUTCOMES:
Transperineal ultrasound measures | 6 months
  Transperineal ultrasound (Voluson E8 Expert from GE Healthcare with a convex RM6C probe ranging from 2 to 6 Megahertz) will be used to measure the function of the pelvic floor muscles indirectly through morphometry at rest, valsalva and at maximum contraction. This imaging will measure the position of the bladder neck relative to the pubis, the anorectal angle formed by the anus and rectum, the angle formed by the pelvic floor muscles and a horizontal reference line (parallel to the ground ) in addition to the dimensions of the urogenital hiatus which is delimited by the puborectal muscle and which includes the urethra, the vagina and the anus. This method has been evaluated in several studies and demonstrates good intra- and inter-rater fidelity
Perineometer measurements | 6 months
  Before starting the assessments as suggested by the International Continence Society, the physiotherapist will check via vaginal palpation the participant's ability to contract and relax the pelvic floor muscles. Afterwords, pelvic examination vaginal manometry (using a Peritron perineometer; Cadio Design, Australia) will be performed to measure resting and maximum contraction of the PFMs

SECONDARY OUTCOMES:
Pelvic floor muscle tenderness scale | 6 months
  Tenderness of each of the PFMs (pubococcygeus, iliococcygeus, coccygeus, and obturator internus muscles) was assessed using a nonvalidated scale from 0 to 4 (0, no pressure or pain; 1, pressure but no pain; 2, pressure with discomfort; 3, moderate pain intensified with muscle contraction; 4, severe pain or inability to perform muscle contraction because of pain). Manometry and the tenderness assessments will be repeated after 60 minutes from the first assessments

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sakıncı, Assos.Prof., Study Chair — Akdeniz University
Locations (1):
- Alime Buyuk, Antalya, Turkey (Türkiye)

REFERENCES:
- [Result] Stuge B, Saetre K, Braekken IH. The association between pelvic floor muscle function and pelvic girdle pain--a matched case control 3D ultrasound study. Man Ther. 2012 Apr;17(2):150-6. doi: 10.1016/j.math.2011.12.004. Epub 2012 Jan 15. PMID 22245422
- [Result] Thibault-Gagnon S, Goldfinger C, Pukall C, Chamberlain S, McLean L. Relationships Between 3-Dimensional Transperineal Ultrasound Imaging and Digital Intravaginal Palpation Assessments of the Pelvic Floor Muscles in Women With and Without Provoked Vestibulodynia. J Sex Med. 2018 Mar;15(3):346-360. doi: 10.1016/j.jsxm.2017.12.017. PMID 29502982